CLINICAL TRIAL: NCT06656598
Title: A Multicenter Randomized Open Label Phase II Study Evaluating the Efficacy and the Tolerance of Immunochemotherapy and of Sequential Hypofractionated Radiotherapy in Unfit or Elderly Patients With Unresectable Stage III Non Small Cell Lung Cancer
Brief Title: Adjuvant Chemotherapy +/- Cemiplimab and Sequential Hypofractionated Radiotherapy in Unfit or Elderly Patients With Stage III Lung Cancer
Acronym: SPORADIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-2401
Record Dates: First submitted 2024-10-09; First posted 2024-10-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Stage III NSCLC
Keywords: NSCLC; NSCLC, Stage III; Unfit or elderly patients; IFCT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; cemiplimab; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (neoadjuvant chemotherapy only) (Active Comparator): Patients will receive neoadjuvant chemotherapy alone with carboplatin AUC 5 D1 and paclitaxel 80mg/m² D1 D8 D15 (3 cycles of 4 weeks). Patients will subsequently receive curative hypofractionated radiotherapy (55 Gy/20fr). After radiotherapy, patients will receive maintenance immunotherapy with Cemiplimab 350 mg every 3 weeks for a period of 12 months.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: Curative hypofractionated radiotherapy; Drug: Cemiplimab (maintenance)
- Arm B (neoadjuvant chemo-immunotherapy) (Experimental): Patients will receive neoadjuvant chemotherapy alone with carboplatin AUC 5 D1 and paclitaxel 80mg/m² D1 D8 D15 and cemiplimab 350 mg D1-D21 (3 cycles of 4 weeks). Patients will subsequently receive curative hypofractionated radiotherapy (55 Gy/20fr). After radiotherapy, patients will receive maintenance immunotherapy with Cemiplimab 350 mg every 3 weeks for a period of 12 months.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Cemiplimab; Radiation: Curative hypofractionated radiotherapy; Drug: Cemiplimab (maintenance)

INTERVENTIONS:
Drug: Carboplatin — Neoadjuvant treatment with Carboplatin AUC 5 D1 (3 cycles of 4 weeks).
Drug: Paclitaxel — Neoadjuvant treatment with Paclitaxel 80mg/m² D1 (3 cycles of 4 weeks).
Drug: Cemiplimab — Neoadjuvant treatment with Cemiplimab (Libtayo®) 350 mg D1-D21 (3 cycles of 4 weeks).
  Arms: Arm B (neoadjuvant chemo-immunotherapy)
Radiation: Curative hypofractionated radiotherapy — Curative hypofractionated radiotherapy (55 Gy/20fr) after the end of neoadjuvant treatment.
Drug: Cemiplimab (maintenance) — Maintenance immunotherapy with Cemiplimab 350 mg every 3 weeks after the end of radiotherapy (12 months).

SUMMARY:
The use of neoadjuvant immuno-chemotherapy could improve survival outcomes of patients eligible for sequential radio-chemotherapy comparing to the benefit already obtained with maintenance immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.
2. Patients must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.
3. Age ≥ 18 years.
4. Histologically or cytologically confirmed locally advanced non small cell lung cancer (NSCLC) stage IIIA non resectable, IIIB or IIIC accordingly to 8th classification TNM, UICC 2015.
5. Patients over 70 years of age with Eastern Cooperative Oncology Group Performance Status (ECOG PS) PS of 0 to 1.

   Or Patients under 70 years of age with ECOG PS of 0 to 1 and a score ≥ 3 according to the Charlson comorbidity criterion or ECOG PS 2.
6. Patients eligible for treatment with sequential radio-chemotherapy validated by multidisciplinary committee.
7. Measurable disease according to RECIST 1.1.
8. Respiratory function:

   * FEV1 ≥ 40% of theoretical value,
   * DLCO ≥ 40%.
9. Bone marrow function:

   * absolute neutrophil count (ANC) ≥ 1.5.109/L,
   * platelets ≥ 100.109/L,
   * hemoglobin ≥ 9 g/dl.
10. Renal and hepatic function:

    * estimated creatinine clearance ≥ 45 ml/min,
    * bilirubin ≤1.5xULN,
    * AST ALT ≤3xULN,
    * Albumin ≥28g/dl.
11. Participant has national health insurance coverage.
12. Effective method of contraception during the treatment and during the 6 months following the last dose for patients of childbearing potential and for male subjects who are sexually active with a woman of childbearing potential.

Exclusion Criteria:

1. Immunotherapy or chemotherapy contra-indicated.
2. Patients eligible for treatment with concomitant radio-chemotherapy validated by multidisciplinary committee.
3. Stage I or II NSCLC.
4. Previously received a treatment with anti-PD1/PDL1, anti-CTLA, or other antineoplastic immunotherapy or chemotherapy for NSCLC.
5. Histology other than primary non-small cell lung cancer.
6. Patients with an activating EGFR mutation or ALK or ROS1 translocation.
7. Metastatic NSCLC including brain metastasis.
8. Patients not eligible for curative radiotherapy (tumor extension, predictable dose constraints that cannot be met).
9. Severe uncontrolled comorbidities or severe intercurrent disease: acute coronary syndrome less than 3 months old, unstable angina, heart failure with LVEF ≤30%, uncontrolled hypertension, Child B or C cirrhosis, severe sepsis, myocarditis or any other active conditions that would contraindicate chemotherapy, immunotherapy, or radiotherapy in the opinion of the investigator.
10. Weight loss ≥15% of total body weight in the last 6 months.
11. ECOG PS upper 2
12. Active autoimmune pathology. History of autoimmune pathology including myasthenia, Guillain-Barre syndrome, lupus erythematosus, antiphospholipid syndrome, Wegener's granulomatosis, glomerulonephritis, inflammatory bowel disease, vasculitis, sarcoidosis, uveitis. Autoimmune thyroid pathologies under replacement therapy as well as type 1 diabetes under insulin are authorized.
13. History of idiopathic pulmonary fibrosis, organized pneumopathy or signs of active interstitial pulmonary pathology on CT scan.
14. Any immunosuppressive therapy received within 28 days and corticosteroids > 10mg/day of prednisone or equivalent received within 7 days prior the start of chemotherapy excepted hydrocortisone replacement for adrenal insufficiency or pituitary disease not considered immunosuppressive therapy.
15. Chronic active infection including tuberculosis, HIV, hepatitis B (HBsAg positive) or C. Patients with a history of cured hepatitis B (anti HBc and absence of negative HBs antigen) are eligible. In case of hepatitis C (anti HCV Ac) patients are eligible if the HCV PCR is negative.
16. Severe infections (including covid-19 infection) within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
17. History of neoplastic disease less than 3 years old or progressive (except basal cell carcinoma of the skin and carcinoma in situ of the uterus).
18. History of thoracic radiotherapy.
19. Live attenuated vaccine received within 28 days of starting chemotherapy
20. History of organ or bone marrow transplantation.
21. Major surgery within 4 weeks of starting treatment.
22. Patient already included in another therapeutic trial.
23. Positive pregnancy test or breastfeeding woman.
24. Protected adults (under guardianship or curatorship).
25. Inability to undergo medical monitoring of the study (for geographical, social and/or physical reasons).
26. Patients unable to understand the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | About 18 months
  Time from randomization to progression or death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | About 18 months
  Proportion of patients who have achieved a best overall response of complete response (CR) or partial response (PR)
Disease Control Rate (DCR) | About 18 months
  Proportion of patients who have achieved a best overall response of complete response (CR) or partial response (PR) or stable disease (SD)
PFS at 12 months | At 12 months
  Time from randomization to progression or death.
PFS at 18 months | At 18 months
  Time from randomization to progression or death.
PFS at 3 year | At 3 year
  Time from randomization to progression or death.
Overall Survival (OS) curve | About 3 year
  Time from date of inclusion to the date of death due to any cause.
OS at 12 months | At 12 months
  Time from date of inclusion to the date of death due to any cause.
OS at 18 months | At 18 months
  Time from date of inclusion to the date of death due to any cause.
OS at 3 year | At 3 year
  Time from date of inclusion to the date of death due to any cause.
Acute and late grade 3-4 toxicity rates of neoadjuvant chemoimmunotherapy before hypofractionated radiotherapy | Up to 90 days after the end of immunotherapy
  Acute and late grade 3-4 toxicity rates by treatment arm according to CTCAE v5.0 up to 90 days after the end of immunotherapy.
To evaluate the quality of life of patients receiving neoadjuvant chemoimmunotherapy before hypofractionated radiotherapy with questionnaire EORTC Quality of Life Questionnaire - Core C30 (QLQ-C30) | About 18 months
  Time to symptom deterioration will be defined as the time from inclusion until the date of first clinically meaningful symptom deterioration (an increase in the score from baseline of ≥10) or death (by any cause) in the absence of a clinically meaningful symptom deterioration, regardless of whether the subject withdraws from therapy or receives another anticancer therapy prior to symptom deterioration.
  The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core Questionnaire C30 (EORTC QLQ-C30) is a 30 item instrument meant to assess some of the different aspects that define the quality of life of cancer patients.
  Scale : Not at all / A little / Quite a bit / Very much
To evaluate the quality of life of patients receiving neoadjuvant chemoimmunotherapy before hypofractionated radiotherapy with questionnaire EORTC Quality of Life Questionnaire - Lung Cancer LC29 (QLQ-LC29). | About 18 months
  Time to symptom deterioration will be defined as the time from inclusion until the date of first clinically meaningful symptom deterioration (an increase in the score from baseline of ≥10) or death (by any cause) in the absence of a clinically meaningful symptom deterioration, regardless of whether the subject withdraws from therapy or receives another anticancer therapy prior to symptom deterioration.
  The EORTC QLQ-LC29 incorporates 5 multi-item scales to assess symptom or quality of life issues.
  Scale : Not at all / A little / Quite a bit / Very much

CONTACTS AND LOCATIONS:
Locations (25):
- France (25):
  - Angers - Centre Paul Papin, Angers
  - Angers - CHU, Angers
  - Avignon - CH, Avignon
  - Boulogne - Ambroise Paré, Boulogne
  - Brest - CHU, Brest
  - Caen - CHU, Caen
  - Caen - CRLCC, Caen
  - Créteil - CHI, Créteil
  - Dijon - CRLCC, Dijon
  - Le Mans - CHG, Le Mans
  - Lille - CRLCC, Lille
  - Marseille - APHM, Marseille
  - Mulhouse - GHRMSA, Mulhouse
  - Paris - Bichat, Paris
  - Paris - Hôpital Cochin, Paris
  - Paris - Tenon, Paris
  - Bordeaux - CHU, Pessac
  - Lyon - HCL, Pierre-Bénite
  - Rennes - CHU, Rennes
  - Rouen - Centre Henri Becquerel, Rouen
  - Nantes - CRLCC, Saint-Herblain
  - Strasbourg - CRLCC, Strasbourg
  - Toulouse - CHU, Toulouse
  - Tours - CHU, Tours
  - Vandoeuvre-lès-Nancy - CRLCC, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided